CLINICAL TRIAL: NCT03997851
Title: Topical Acetaminophen for Itch Relief: a Proof of Concept Study in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gil Yosipovitch, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20190133
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Acetaminophen; carbomer

STUDY DESIGN:
Intervention Model Description: The antipruritic effect of 3 topical treatments of varying doses and 1 vehicle treatment will be explored in each subject. One study visit will consist of testing all topical formulations on histaminergic induced itch, and second study visit will test all topical formulations on non-histaminergic induced itch.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Topical 5% acetaminophen gel (Experimental): Topical 5% acetaminophen gel will be applied to one 4x4 cm predefined skin area on the ventral forearm during 2 study visits. The gel will be applied to the test area and will be allowed 30 minutes to adsorb. Following this pre-treatment, residual gel will be removed and itch induction/sensory testing will commence, strictly within the pre-treated area.
  Interventions: Drug: Acetaminophen
- Topical 2.5% acetaminophen gel (Experimental): Topical 2.5% acetaminophen gel will be applied to one 4x4 cm predefined skin area on the ventral forearm during 2 study visits. The gel will be applied to the test area and will be allowed 30 minutes to adsorb. Following this pre-treatment, residual gel will be removed and itch induction/sensory testing will commence, strictly within the pre-treated area.
  Interventions: Drug: Acetaminophen
- Topical 1% acetaminophen gel (Experimental): Topical 1% acetaminophen gel will be applied to one 4x4 cm predefined skin area on the ventral forearm during 2 study visits. The gel will be applied to the test area and will be allowed 30 minutes to adsorb. Following this pre-treatment, residual gel will be removed and itch induction/sensory testing will commence, strictly within the pre-treated area.
  Interventions: Drug: Acetaminophen
- Topical vehicle gel (Placebo Comparator): Topical vehile gel will be applied to one 4x4 cm predefined skin area on the ventral forearm during 2 study visits. The gel will be applied to the test area and will be allowed 30 minutes to adsorb. Following this pre-treatment, residual gel will be removed and itch induction/sensory testing will commence, strictly within the pre-treated area.
  Interventions: Drug: Carbomer 980

INTERVENTIONS:
Drug: Acetaminophen — Topical acetaminophen gel
  Other Names: Topical acetaminophen gel
  Arms: Topical 1% acetaminophen gel; Topical 2.5% acetaminophen gel; Topical 5% acetaminophen gel
Drug: Carbomer 980 — Topical vehicle gel
  Other Names: Topical vehicle gel
  Arms: Topical vehicle gel

SUMMARY:
Currently, topical antihistamines and corticosteroids are mainly used for itching relief. However, the over the counter antihistamines are not effective on all itch conditions. Acetaminophen is a popular and widely used OTC drug for pain relief. Although its mode of action is still unknown, recent studies have shown that acetaminophen indirectly activates cannabinoid CB1 receptors. Recent studies have shown that topical cannabinoid agonists are effective for itch relief, the efficacy of topical acetaminophen will be tested for non-histaminergic itch relief.

DETAILED DESCRIPTION:
This will be a single-blinded, vehicle-controlled randomized study in healthy controls to test the efficacy of the topical gel formulation with three differing concentrations of acetaminophen (APAP) for itch relief. To detect medium effects of the treatments with a given α of 0.5 and an error probability of 0.05, with a power of 0.95, the number of participants needed is 36 (10 within post hoc pairwise comparisons).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects must be between 18 and 50 years of age.
2. Must be in general good health with no disease or physical conditions that would impair evaluation of itch and pain perception.
3. No history of chronic itch or pain.
4. Must abstain from the use of any systemic or topical anti-histamine, steroid, or pain relief medications from the week prior to the study till the completion of the study.
5. Must abstain from the use of moisturizers on the arms 24 hours before study visits.

Exclusion Criteria:

1. Individuals under 18 or over 50 years of age.
2. Inability to complete the required measures.
3. The presence of an itchy skin disease.
4. Diagnosis of diseased that would affect itch or pain perception (e.g. neuropathies).
5. Currently enrolled in any investigational study in which the subject is receiving any type of drug, biological, or non-drug therapy.
6. Use of oral, topical analgesics, or other medications known to interfere with itch or pain perception in the week prior to the study and throughout the study (e.g. antihistamines, anesthetics, opioids, neuroleptics, etc.).
7. Use of emollients on the arms a week prior to the study and throughout the study.
8. Known allergies to acetaminophen and cowhage.
9. Pregnant women. (Women of child bearing potential will undergo an hCG pregnancy test).
10. Currently incarcerated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: skin arm test areas
Groups:
- Topical acetaminophen and vehicle gel: Each participant will receive topical gel treatments applied for 30 minutes to 4 separate 4 x 4 cm predefined skin areas on the ventral forearms twice at 2 separate study visits.
  The 4 treatments are:
  5% acetaminophen gel 2.5% acetaminophen gel
  1% acetaminophen gel Vehicle gel
  Acetaminophen: Topical acetaminophen gel
Period: Overall Study
Arm/Group | Topical acetaminophen and vehicle gel
Started | 17; 136 skin arm test areas
Completed | 17; 136 skin arm test areas
Not Completed | 0; 0 skin arm test areas

BASELINE CHARACTERISTICS:
Population: Each participant will receive 4 topical gel treatments twice at 2 separate study visits.
  The 4 treatments are:
  5% acetaminophen gel 2.5% acetaminophen gel
  1% acetaminophen gel Vehicle gel
  Acetaminophen: Topical acetaminophen gel
Arm/Group | Topical Acetaminophen and Vehicle Gel
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Itch Intensity Between the Vehicle and Active Treatments During Non-histaminergic Itch Induction
Description: Peak itch intensity between the vehicle and 3 other active treatments (5%, 2.5%, and 1% acetaminophen gels) after non-histaminergic itch induction (cowhage). Itch intensity was measured on a 10cm scale visual analog scale for 10 minutes. 0 was weighted with "no itch" and 10 was weighted with "most itch imaginable".
Time Frame: 10 minutes
Population: All subjects received 4 topical cream treatments.
Measure: Mean (Standard Deviation); unit: Intensity score
Arm/Group | Topical 5% acetaminophen gel | Topical 2.5% acetaminophen gel | Topical 1% acetaminophen gel | Topical vehicle gel
Number analyzed (Participants) | 17 | 17 | 17 | 17
Intensity score | 4.5 (1.98) | 3.94 (2.77) | 5.32 (2.29) | 5.79 (2.61)

2. Primary Outcome: Peak Itch Intensity Between the Vehicle and Active Treatments During Histaminergic Itch Induction
Description: Peak itch intensity between the vehicle and 3 other active treatments (5%, 2.5%, and 1% acetaminophen gels) after histaminergic itch induction. Itch intensity was measured on a 10cm scale visual analog scale for 10 minutes. 0 was weighted with "no itch" and 10 was weighted with "most itch imaginable".
Time Frame: 10 minutes
Population: All subjects received 4 topical cream treatments.
Measure: Mean (Standard Deviation); unit: Intensity score
Arm/Group | Topical 5% acetaminophen gel | Topical 2.5% acetaminophen gel | Topical 1% acetaminophen gel | Topical vehicle gel
Number analyzed (Participants) | 17 | 17 | 17 | 17
Intensity score | 2.04 (2.52) | 2.38 (2.26) | 2.91 (2.31) | 3.07 (2.64)

3. Secondary Outcome: Thermal Threshold Detection (Heat Pain)
Description: Standardized quantitative sensory testing is performed to measure heat pain threshold (assesses the threshold at which heat pain sensation is first detected). Measured in Celsius.
Time Frame: 3 minutes
Population: All subjects received treatment with the 4 topical cream formulations at 2 study visits. Quantitative sensory testing was performed on each area of treated skin.
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Topical 5% acetaminophen gel | Topical 2.5% acetaminophen gel | Topical 1% acetaminophen gel | Topical vehicle gel
Number analyzed (Participants) | 17 | 17 | 17 | 17
Degrees celsius
  After histamine itch induction | 43.95 (2.17) | 44.51 (0.72) | 43.94 (0.88) | 44.07 (0.56)
  After non-histamine itch induction | 43.99 (0.95) | 44.03 (0.81) | 44.30 (0.64) | 44.20 (0.59)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks.
Arm/Group | Topical 5% acetaminophen gel | Topical 2.5% acetaminophen gel | Topical 1% acetaminophen gel | Topical vehicle gel
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03997851/Prot_SAP_000.pdf